CLINICAL TRIAL: NCT03761992
Title: Measurement of the Effect of Gingko Biloba Extract on Ocular and Nailfold Blood-flow in Normaltension Glaucoma by Ocular Coherence Tomography Angiography and Nailfold Capillaroscopy
Brief Title: Measurement of the Effect of Gingko Biloba Extract on Ocular and Nailfold Blood-flow in NTG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Robert Ritch, MD, LLC. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFC Gingko
Record Dates: First submitted 2018-11-20; First posted 2018-12-03 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Normal Tension Glaucoma
MeSH Terms: conditions — Low Tension Glaucoma

STUDY DESIGN:
Intervention Model Description: Gingko baloba extract (GBE) versus placebo
Who Masked: Participant, Investigator
Masking Description: Neither the patient nor the investigator will know which treatment that the patient is receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gingko Biloba Extract (Active Comparator): Gingko Biloba Extract 240 mg.
  Interventions: Dietary Supplement: Gingko Baloba
- Placebo (Placebo Comparator): Placebo Pill
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Gingko Baloba — Tablets
  Other Names: 240mg. Gingko Biloba
  Arms: Gingko Biloba Extract
Other: Placebo — Tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of Ginkgo biloba extract (GBE) on the number of blood vessels in the back of the eye as well as the amount of blood flow at the nailfold(where the fingernail meets the skin) of the 4th finger in the hand.This finger, along with the 5th finger, has the most transparent skin, which makes imaging a little easier. GBE is an over-the-counter pill, made from a natural powder taken from the Gingko (Maidenhair) tree, that is widely used. A technique called Optical Coherence Tomography Angiography (OCTA),will be used to measure the small blood vessels at the back of the eye, the macula (the area of sharpest vision), and the optic disc (the point at which the nerve fibers from the retina enter to form the optic nerve, which transmits visual impulses to the brain).

DETAILED DESCRIPTION:
GBE has been reported to improve blood flow to the brain, eye, and extremeties(hands, feet,etc.). .As with most supplements, GBE is neither regulated nor FDA approved.

A technique called Optical Coherence Tomography Angiography (OCTA),will be used to measure the small blood vessels at the back of the eye, the macula (the area of sharpest vision), and the optic disc (the point at which the nerve fibers from the retina enter to form the optic nerve, which transmits visual impulses to the brain). This technique uses a camera, capable of imaging the smallest vessels, so that their density (number) can be calculated by a computer. This is being done to determine if there is disease causing increasing loss of these vessels. The imaging is done by a widely used camera which does not contact the eye. It simply uses visible light to measure the amount of blood vessels present in a determined area in the back of the eye. Blood flow at the 4th finger nailfold (nailfold capillaroscopy; NFC) is a standard technique, especially in rheumatology, performed by using a commercially available light microscope which glides over the base of the fingernail and can image the tiny capillaries in the nailfold. These images are recorded as videos from which the blood flow can be analyzed by freely available software for the purpose of quantitative measurements (amount of blood flow and blood flow velocity).

ELIGIBILITY:
Inclusion Criteria:

Male or female of any race, at least 18 years of age

* Has provided verbal and written informed consent.
* Able and willing to follow instructions, including participation in all study assessments and visits.
* Eyes with NTG will be enrolled.
* Glaucoma severity will be graded using the WHO (World Health Organization)staging system.

NTG diagnosis will be based on the following:

1. Glaucomatous optic disc on slit-lamp biomicroscopy defined as cup-to-disc ratio greater than 0.7, inter-eye asymmetry in cup-to-disc ration greater than 0.2 or neuroretinal rim notching, focal thinning, disc hemorrhage or vertical elongation of optic disc.
2. Glaucomatous visual field defects on at least three reliable visual field examinations as measured by a glaucoma hemifield test (GHT) result outside normal limits and/or the appearance of at least three consecutive test points on the pattern deviation plot with p<1% and at least one at p<0.05%, not including points on the edge of the field.
3. NTG will be defined as those subjects with a history of untreated peak IOP ≤21 mmHg.

   * Both eyes will be enrolled

Exclusion Criteria:

* Best-corrected visual acuity less than 20/40
* Age younger than 18 years or older than 85 years
* Refractive error greater than +3.00 diopters (D) or less than -7.00 diopters (D)
* Previous intraocular surgery except for uncomplicated cataract extraction with posterior chamber intraocular lens implantation
* Any other diseases that may cause visual field loss or optic disc abnormalities
* Inability to perform reliably on automated visual field testing.
* Subjects taking any GBE product will be washed out for 2 weeks prior to enrollment.
* Diabetes.
* Seizure disorder.
* Taking any drugs that may interact with GBE (as listed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome - Measure of Blood Vessel by Optical Cohrence Tomography Angiography (OCTA) | 4 weeks
  The investigators plan to evaluate the density of the small blood vessels at the back of the eye. This will be measured by a OCTA. A camera capable of imaging the smallest vessels so that their density (number) can be calculated by a computer, the purpose being to determine if there is disease causing progressive loss of these vessels.

SECONDARY OUTCOMES:
Secondary Outcome - Measure of Blood Flow and Velocity by Nailfold Capillaroscopy (NFC) | 4 weeks
  Measuring blood flow at the 4th finger nailfold by NFC is a standard technique, especially in rheumatology, in which a commercially available light microscope glides over the base of the fingernail to image the tiny capillaries in the nailfold. These images are recorded as videos from which the blood flow can be analyzed quantitatively by freely available software to measure blood flow and velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ritch, MD, Principal Investigator — New York Eye and Ear Infirmary of mount Sinai
Locations (1):
- New York Eye and Ear Infirmary of Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940
- [Background] Kim KE, Park KH. Update on the Prevalence, Etiology, Diagnosis, and Monitoring of Normal-Tension Glaucoma. Asia Pac J Ophthalmol (Phila). 2016 Jan-Feb;5(1):23-31. doi: 10.1097/APO.0000000000000177. PMID 26886116
- [Background] Pasquale LR. Vascular and autonomic dysregulation in primary open-angle glaucoma. Curr Opin Ophthalmol. 2016 Mar;27(2):94-101. doi: 10.1097/ICU.0000000000000245. PMID 26720776
- [Background] Flammer J, Konieczka K, Flammer AJ. The primary vascular dysregulation syndrome: implications for eye diseases. EPMA J. 2013 Jun 7;4(1):14. doi: 10.1186/1878-5085-4-14. PMID 23742177